CLINICAL TRIAL: NCT01485380
Title: Combined Electroencephalogram, Magnetic Resonance Imaging-Positron Emission Tomography of Dexmedetomidine Induced Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Assistant in Anesthaesia, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-P-002333
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Dexmedetomidine Induced Sedation
Keywords: Dexmedetomidine; Sleep; MRI-PET; EEG
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active study arm (Experimental): Subjects recruited into this study will be required to undergo two magnetic resonance imaging- positron emission tomography (MRI-PET) scans of the brain in addition to high density electroencephalogram (EEG) acquisition. The first scan will be a baseline scan while the second scan will be performed while dexmedetomidine is being infused.
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — The dexmedetomidine infusion will be individualized to each study participant by a target plasma concentration where loss of consciousness is initially observed. Loss of consciousness will be assayed by specific auditory and verbal stimuli.
  Other Names: precedex

SUMMARY:
The investigators are doing this research study to find out how and where dexmedetomidine, a sedative anesthetic, acts in the brain. The investigators will do this by using a machine that records the brains electrical activity, called an electroencephalogram (EEG), and brain imaging scans to look at the brain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I
* 18 to 35 years of age

Exclusion Criteria:

* MRI and/or PET screening criteria not met
* Abnormal sleep habits/known or suspected sleep disorder(s)
* Taking medication that alters sleep, cognitive function, or both -History of a known neurological or psychiatric problem -Younger than 18 or older than 35 years of age

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Johnson-Akeju, M.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Study Arm: Subjects recruited into this study will be required to undergo two magnetic resonance imaging-positron emission tomography scans of the brain in addition to high density electroencephalogram acquisition. The first scan will be a baseline scan while the second scan will be performed while dexmedetomidine is being infused.
  dexmedetomidine: The dexmedetomidine infusion will be individualized to each study participant by a target plasma concentration where loss of consciousness is initially observed. Loss of consciousness will be assayed by specific auditory and verbal stimuli.
Period: Overall Study
Arm/Group | Active Study Arm
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Active Study Arm: Subjects recruited into this study will be required to undergo two MRI-PET scans of the brain in addition to high density electroencephalogram acquisition. The first scan will be a baseline scan while the second scan will be performed while dexmedetomidine is being infused.
  dexmedetomidine: The dexmedetomidine infusion will be individualized to each study participant by a target plasma concentration where loss of consciousness is initially observed. Loss of consciousness will be assayed by specific auditory and verbal stimuli.
Arm/Group | Active Study Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in the Brains Default Mode Network.
Description: Number of participants with changes in the Default Mode network during loss and recovery of consciousness under dexmedetomidine induced sedation versus baseline as assessed by changes in blood oxygen level depended (BOLD) signals during the awake, unconscious, and recovery states.
Time Frame: 1.5hrs
Population: All 17 participants were analyzed. Blood oxygen level depended (BOLD) signals during the awake (n = 16), unconscious (n = 16), and recovery (n = 15) states were included in the final data set.
Measure: Number; unit: participants
Groups:
- Active Study Arm: Subjects recruited into this study will be required to undergo two magnetic resonance imaging-positron emission tomography (MRI-PET) scans of the brain in addition to high density electroencephalogram (EEG) acquisition. The first scan will be a baseline scan while the second scan will be performed while dexmedetomidine is being infused.
  dexmedetomidine: The dexmedetomidine infusion will be individualized to each study participant by a target plasma concentration where loss on consciousness is initially observed. Loss on consciousness will be assayed by specific auditory and verbal stimuli.
Arm/Group | Active Study Arm
Number analyzed (Participants) | 17
participants | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire duration of the study.
Description: Adverse events were systematically characterized according to our research protocol.
Groups:
- Active Study Arm: Subjects recruited into this study will be required to undergo two MR-PET scans of the brain in addition to high density EEG acquisition. The first scan will be a baseline scan while the second scan will be performed while dexmedetomidine is being infused.
  dexmedetomidine: The dexmedetomidine infusion will be individualized to each study participant by a target plasma concentration where loss of consciousness is initially observed. Loss of consciousness will be assayed by specific auditory and verbal stimuli.
Arm/Group | Active Study Arm
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes